CLINICAL TRIAL: NCT03036319
Title: Patient-Centered NeuroRehabilitation
Brief Title: Patient-Centered NeuroRehabilitation (PCN)
Acronym: PCN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00111090
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Deficit
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Masking Description: Given the nature of this study, the participant, care provider, investigator, and/or outcome assessors may or may not be blinded to the treatment condition.
Oversight: Data Monitoring Committee: No

ARMS (7):
- Active TES (Experimental): Participants will receive "real" tES (tDCS, tACS, tRNS) in which they receive up to 4 milliamps (mA) of stimulation per electrode for up to 40 minutes for up to 260 sessions. As this may be a cross-over design, some participants may receive active and sham conditions.
  Interventions: Device: Active tDCS; Device: Active tACS; Device: Active tRNS
- Sham TES (Placebo Comparator): Participants undergoing this condition will have the exact same procedures as the active group, with the exception that they will receive only sham stimulation for up to 260 sessions.
  Interventions: Device: Sham tDCS; Device: Sham tACS; Device: Sham tRNS
- Cognitively based intervention (Experimental): Participants may receive a cognitively based intervention that targets the particular cognitive and/or functional abilities of interest. This includes methods of cognitive training, cognitive remediation, and cognitive rehabilitation.
  Interventions: Behavioral: Cognitively based intervention
- Active TES + Cognitively based intervention (Experimental): This condition combines active TES and cognitively based interventions for some or all of the study sessions
  Interventions: Device: Active tDCS; Behavioral: Cognitively based intervention; Device: Active tACS; Device: Active tRNS
- Sham TES + Cognitively based intervention (Experimental): This condition combines sham TES and cognitively based interventions for some or all of the study sessions
  Interventions: Device: Sham tDCS; Behavioral: Cognitively based intervention; Device: Sham tACS; Device: Sham tRNS
- Active TES, Sham TES, Cognitively based interventions (Experimental): This condition combines active and sham TES with cognitively based interventions using a cross-over design
  Interventions: Device: Active tDCS; Device: Sham tDCS; Behavioral: Cognitively based intervention; Device: Active tACS; Device: Sham tACS; Device: Active tRNS; Device: Sham tRNS
- Active and Sham TES (Experimental): Participants will receive active and sham TES
  Interventions: Device: Active tDCS; Device: Sham tDCS; Device: Active tACS; Device: Sham tACS; Device: Active tRNS; Device: Sham tRNS

INTERVENTIONS:
Device: Active tDCS — Participants will receive active tDCS at up to 4mA per electrode for up to 40 minutes for up to 260 sessions.
  Arms: Active TES; Active TES + Cognitively based intervention; Active TES, Sham TES, Cognitively based interventions; Active and Sham TES
Device: Sham tDCS — Participants will receive sham tDCS for up to 260 sessions
  Arms: Active TES, Sham TES, Cognitively based interventions; Active and Sham TES; Sham TES; Sham TES + Cognitively based intervention
Behavioral: Cognitively based intervention — Participants may receive a cognitively based intervention that targets the particular cognitive and/or functional abilities of interest. This includes methods of cognitive training, cognitive remediation, and cognitive rehabilitation for up to 260 sessions
  Arms: Active TES + Cognitively based intervention; Active TES, Sham TES, Cognitively based interventions; Cognitively based intervention; Sham TES + Cognitively based intervention
Device: Active tACS — Participants will receive active transcranial alternating current stimulation at up to 4mA per electrode for up to 40 minutes for up to 260 sessions
  Arms: Active TES; Active TES + Cognitively based intervention; Active TES, Sham TES, Cognitively based interventions; Active and Sham TES
Device: Sham tACS — Participants will receive sham transcranial alternating current stimulation for up to 260 sessions
  Arms: Active TES, Sham TES, Cognitively based interventions; Active and Sham TES; Sham TES; Sham TES + Cognitively based intervention
Device: Active tRNS — Participants will receive active transcranial random noise stimulation at up to 4mA per electrode for up to 40 minutes for up to 260 sessions
  Arms: Active TES; Active TES + Cognitively based intervention; Active TES, Sham TES, Cognitively based interventions; Active and Sham TES
Device: Sham tRNS — Participants will receive sham transcranial random noise stimulation for up to 260 sessions
  Arms: Active TES, Sham TES, Cognitively based interventions; Active and Sham TES; Sham TES; Sham TES + Cognitively based intervention

SUMMARY:
As individuals grow older, a number of factors can reduce our cognitive (or thinking) abilities such as "normal" aging, neurodegenerative diseases, and cardiovascular disease. This study will evaluate whether cognitive rehabilitation and transcranial electrical stimulation (TES) can improve cognitive abilities. Cognitive rehabilitation refers to methods that are used to improve tasks people have trouble doing in everyday life. Transcranial electrical stimulation uses small amounts of electricity to try to alter brain functioning. These approaches may help improve cognitive abilities like attention, learning, memory, finding words, and problem solving as well as everyday functioning. The goal of this study is to identify how to best use these methods, either alone or in combination.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the feasibility of a neurorehabilitation treatment tailored to individual patient needs, with the ultimate goal of maximizing cognitive and real-world functioning for older adults with cognitive aging, mild cognitive impairment (MCI), neurodegenerative, or other neurological diseases/conditions.

Transcranial electrical stimulation (TES) is a non-invasive, neurorehabilitation procedure in which a weak electric current is passed between electrodes that are placed on the scalp with the intention of modulating excitability of the underlying brain regions. Because the field of TES is relatively young, rapidly evolving, and primarily focused on cognitive neuroscience with "healthy" individuals, there is a clear need for well-conceptualized and conducted clinical research. The current protocol is intentionally broad with respect to both methodology and patient characteristics in order to tailor potential TES interventions to individual patients or small samples. The current protocol utilizes various forms of TES including transcranial direct current stimulation (tDCS), alternating current stimulation (tACS), and random noise stimulation (tRNS) and sham stimulation in older adults. As this is a cross-over design, some participants may receive active (or "real") TES and/or sham TES conditions.This includes head to head comparisons of the different forms of TES. Additionally, TES could be performed in conjunction with cognitively-based intervention since this may enhance the neuroplastic response of the targeted brain region(s) while at the same time shaping/optimizing the pathways that are engaged by cognitively-based interventions. This broad approach is important since etiological differences in cognitive impairment may necessitate distinct interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have reported cognitive dysfunction and cognitively intact participants.
2. Participants will be age 50 or older

Exclusion Criteria:

1. A history of epilepsy
2. Sensory or motor impairments that limit the ability to take part in the study
3. Current alcohol or drug abuse/dependence
4. Those who are currently pregnant or may become pregnant during the duration of the study (if there is a question of pregnancy, pregnancy tests will be available for participants at no charge)

Those who are being evaluated for TES methodology will also be excluded for 1) metallic or electronic implant 2) skull plates or other cranial implants that affect TES

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-06; Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
TES side effect questionnaire | Immediately following TES (<15 minutes)
  Side effect questionnaire that asks participants to rate the severity of potential TES related side effects

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Hampstead, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - Department of Psychiatry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No